CLINICAL TRIAL: NCT05022628
Title: Clinical Study of Radiotherapy Combined With Donafenib for Neoadjuvant Treatment of Patients With HCC With Portal Vein Carcinoma Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ky153
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: HCC; Chemotherapy Effect
MeSH Terms: interventions — donafenib; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Therapy arm (Experimental): donafenib
  Interventions: Drug: Donafenib

INTERVENTIONS:
Drug: Donafenib — Donafenib treatment regimen.
  1. Donafenib started on the day of the first radiation treatment.
  2. starting dose 0.2 g bid twice daily orally on an empty stomach (1 hour before or 2 hours after a meal).
  3. Surgery after at least 1 week off Donafinil; resume Donafinil dosing as soon as possible after postoperative wound healing until any of the following occurs, whichever occurs first: (i) the subject develops an intolerable toxic reaction that does not resolve after dose adjustment (see 5.3 for details); (ii) 12 months of postoperative dosing; (iii) the subject has the first imaging-confirmed recurrence of disease or withdraws from the study (whichever occurs first).
  4. Dose adjustment/withdrawal: Subjects are allowed up to 2 dose adjustments if they experience an adverse event related to the trial drug during treatment.
  Other Names: Radiotherapy

SUMMARY:
For HCC patients with combined PVTT, systemic therapy can be used as a basic approach throughout the treatment and in combination with hepatectomy, TACE, HAIC, radiotherapy, etc.

Our center proposes to conduct a clinical study of radiotherapy combined with donafinil for neoadjuvant treatment of HCC patients with portal vein carcinoma thrombosis to observe the safety and efficacy of donafinib combined with radiotherapy for neoadjuvant treatment

Translated with www.DeepL.com/Translator (free version)

DETAILED DESCRIPTION:
In the pre-enrollment screening phase, investigators are required to record all screened patients uniformly on a subject screening and enrollment form that focuses on basic patient information (name, date of birth, and gender), date of screening received, and outcome (e.g., included in the study, not included in the study, and their reasons). The screening items in this phase are all part of the routine clinical treatment process, and the results of the tests performed before the patient signs the informed consent form can be used for evaluation. Patients who subsequently meet all inclusion and exclusion criteria are required to sign the informed consent form before they can be enrolled in the trial.

Patients with hepatocellular carcinoma who meet the inclusion criteria are fully evaluated during the screening phase to see if they meet the enrollment criteria.

Complete the following items within 28 days prior to treatment initiation.

* Obtain a written signed ICF.
* Demographic information: including date of birth, gender, ethnicity/race.
* History of alcohol consumption, history of smoking.
* Past medical and treatment history: take all past medical and treatment histories other than this indication that began prior to signing the ICF and that are considered relevant to this study.
* Physical examination: including head, eyes, ears, nose, throat, neck, heart, chest (including lungs), abdomen, extremities, skin, lymph nodes, nervous system, and general condition of the subject.
* Height and weight measurements.
* Vital signs: temperature, respiration, blood pressure and heart rate.
* ECOG score: it is recommended that the ECOG evaluation be performed by the same investigator throughout the study period, as detailed in Appendix 4.
* Child-Pugh score (Appendix 5).
* CNLC staging and Barcelona liver cancer staging.
* Virological testing: hepatitis B two-for-half [including hepatitis B virus surface antibody (HBsAb), HBsAg, hepatitis B virus e antigen (HBeAg), hepatitis B virus e antibody (HBeAb), and HBcAb], HCV antibody, and HIV antibody.
* Review of inclusion and exclusion criteria to assess the eligibility of subjects for inclusion.
* AE collection: for AEs after signing the ICF and before the first dose, they should be recorded on the past medical history page of the CRF.

Complete the following items within 14 days prior to treatment initiation.

* Routine blood tests including: red blood cell count, hemoglobin, red blood cell pressure, white blood cell count and classification (neutrophils, lymphocytes, eosinophils, monocytes, basophils), and platelet count; obtain baseline values within 14 days prior to enrollment.
* Blood biochemical tests including: total protein, albumin, creatinine, ALP, lactate dehydrogenase, total bilirubin, direct bilirubin, AST, ALT, calcium, phosphorus, potassium, sodium, and chloride.
* Routine urine examination including: specific gravity, pH, urine sugar, protein, tubular, ketone bodies, blood cells; 24-hour urine protein quantification is required if 2 consecutive urine protein tests are ++ or more or if the physician judges the results to be abnormal and clinically significant.
* Fecal occult blood
* Coagulation tests including: aPTT, PT, TT, INR
* Blood pregnancy test: female subjects of childbearing age only.
* 12-lead electrocardiogram (ECG).
* alpha-fetoprotein (AFP).
* HBV-DNA quantification: HBV-infected subjects only.
* Tumor assessment: screening tumor assessment must be performed within 14 days prior to enrollment and should include a CT or MRI scan of the chest, abdomen, or pelvis; if clinically indicated, any other known or suspected disease site may be examined using appropriate methods, such as a cranial MRI, bone scan, or CT scan of the neck; imaging of tumors done for routine visits before the subject signs up for ICF need not be repeated if done within 3 weeks prior to enrollment and at this study center; baseline and follow-up assessments should be performed using the same imaging methods and assessed by the same investigator whenever possible.
* Combined medication/combined treatment collection: all medication received by the subject from 14 days prior to enrollment must be recorded in the CRF, including the generic name and daily dose of the medication, the reason for the use of that medication, the start date and the end date.
* Assign enrollment number.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 75 years (inclusive of cut-offs), male or female. Histologically confirmed HCC or meeting the AASLD guidelines for clinical diagnostic criteria for HCC.

Patients with primary HCC without prior systemic therapy (except antiviral therapy) or local therapy and at least 1 measurable lesion meeting the definition of mRECIST criteria.

Chinese primary liver cancer staging (CNLC) IIIa, Cheng's portal PVTT staging type II/III, tumor confined to a single liver lobe, tumor load <50%.

Liver function Child-Pugh score of 5-7. Eastern Cooperative Oncology Group (ECOG) physical status (PS) score 0-1. Expected survival of not less than 3 months. HBV-infected patients with HBV-DNA of ≥104copies/ml within 14 days prior to enrollment, followed by antiviral therapy (entecavir recommended) down to <104copies/ml before study entry, and continued antiviral therapy and monitoring of liver function and serum HBV-DNA levels.

Have adequate organ function reserve and laboratory test values within 14 days prior to treatment must meet the following criteria.

Routine blood tests. Hb≥100 g/L ANC ≥ 1.5×109 /L PLT ≥ 75×109 /L Biochemical examination. ALB ≥28g/L ALT and AST <5×ULN TBIL ≤1.5×ULN Creatinine ≤1.5×ULN or creatinine clearance (Ccr) ≥50 mL/min Creatinine clearance needs to be calculated by the Cockcroft-Gault formula. Men. Creatinine clearance = ((140 age) × body weight (kg))/(72 × serum creatinine (mg/dL)) Females: Male calculation × 0.85. Basic normal electrolytes or normal with treatment. Urine protein <2+ or quantitative 24-hour urine protein test ≤1.0 g/L (for patients with urine protein ≥2+, quantitative 24-hour urine protein test must be ≤1.0 g/L to be enrolled).

Coagulation function. International standard ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN Activated partial clotting time (aPTT) ≤ 1.5 x ULN Patients were voluntarily enrolled, able to provide written informed consent, and able to understand and comply with the trial protocol for medication administration and follow-up.

Exclusion Criteria:

* Pre-existing or co-morbidities.

  1. pathologically confirmed hepatocellular carcinoma-intrahepatic cholangiocarcinoma (HCC-ICC) mixed or fibrous lamellar-like hepatocellular carcinoma.
  2. recurrent hepatocellular carcinoma.
  3. previous local treatment (including hepatectomy, liver transplantation, TACE, HAIC, radiotherapy, etc.) or systemic treatment (except antiviral therapy)
  4. multiple (number of nodules >3) or diffuse intrahepatic nodules
  5. presence of inferior vena cava carcinoma thrombosis, hepatic vein carcinoma thrombosis or bile duct carcinoma thrombosis, extrahepatic metastases or tumor load >50%.
  6. the presence of other malignancies within 5 years, unless the patient has received potentially curative treatment and there has been no evidence of the presence of that disease within 5 years, except that this time requirement (i.e., within 5 years) does not apply to patients with successfully resected basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, or other carcinoma in situ
  7. A prior history of serious psychiatric illness.
  8. medical conditions affecting the absorption, distribution, metabolism or clearance of the study drug (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorders, etc.) Pre-existing or combined medication/treatment.
  9. Have undergone major surgery (as determined by the investigator) within 4 weeks prior to enrollment.
  10. Patients who have received other systemic antitumor therapy prior to enrollment, including other herbal medicines with antitumor indications, for less than 2 weeks or 5 drug half-lives (whichever is longer) after completion of treatment until dosing in this study, or who have not recovered to ≤ CTCAE grade 1 from adverse events caused by preoperative therapy.
  11. Concomitant administration of drugs that may prolong QTc and/or induce tip-twisting ventricular tachycardia (Tdp) or that affect drug metabolism.

      Safety.
  12. Patients with a known or suspected history of allergy to tyrosine kinase inhibitor (TKI) drugs or to excipients of the study drug.
  13. Presence of uncontrollable hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion or pericardial effusion.
  14. presence of active bleeding or coagulation abnormalities, bleeding tendency or being treated with thrombolytic, anticoagulant or antiplatelet therapy
  15. history of gastrointestinal bleeding within the previous 4 weeks or a definite propensity for gastrointestinal bleeding (e.g., known localized active ulcer lesions, fecal occult blood ++, gastroscopy if persistent fecal occult blood +), or other conditions that may cause gastrointestinal bleeding as determined by the investigator (e.g., severe fundic/esophageal varices).
  16. Gastrointestinal perforation, abdominal fistula or abdominal abscess within the previous 6 months
  17. thrombosis or thromboembolic event within the previous 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc.
  18. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina or coronary artery bypass grafting within the previous 6 months, congestive heart failure (New York Heart Association NYHA class >2), arrhythmias that are poorly controlled or require pacemaker therapy, hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg) that is not controlled by medication.
  19. Active infection, including. Positive for HIV (HIV) (HIV1/2 antibodies). Active hepatitis C (positive HCV antibodies or HCV-RNA ≥ 103 copies/ml and abnormal liver function).

      Active co-infection with hepatitis B virus (HBV) and hepatitis C virus (HCV). Active tuberculosis. Other uncontrollable active infections (CTCAE V5.0 > grade 2).
  20. Other significant clinical and laboratory abnormalities that, in the opinion of the investigator, affect the safety evaluation, e.g., uncontrolled diabetes mellitus, chronic kidney disease, grade II or higher peripheral neuropathy (CTCAE V5.0), abnormal thyroid function, etc.
  21. Pregnant or lactating women, and female or male patients of childbearing potential who are unwilling or unable to use effective contraception.

      Other.
  22. History of alcohol, psychotropic or other substance abuse within the previous 6 months.
  23. having received another drug or medical device clinical trial within 4 weeks prior to enrollment
  24. Inability to follow the study protocol for treatment or scheduled follow-up.
  25. Any other person who, in the opinion of the investigator, cannot be enrolled in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | 2 years
  The incidence of adverse-effect and severe adverse-effect

IPD SHARING:
Plan to Share IPD: Undecided